CLINICAL TRIAL: NCT03836755
Title: Evaluation of the Stability of Osseointegrated Implant in Upper Limb or Lower Limb Amputees
Brief Title: Evaluation of the Stability of Osseointegrated Implant in Amputees
Acronym: METACOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other); Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other); Scuola Universitaria Superiore Sant'Anna Pisa (Unknown)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor and Head of department, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 33/18
Record Dates: First submitted 2019-02-05; First posted 2019-02-11 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Prosthesis Migration; Amputation
Keywords: osseointegration; implant migration; amputee
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- METACOS (Other): Required to do some motor tasks during static and dynamic RSA
  Interventions: Diagnostic Test: Metacos

INTERVENTIONS:
Diagnostic Test: Metacos — Evaluation of stability of implant by RSA technique

SUMMARY:
The study concerns the technique of osseointegration that consists of inserting a titanium pin into the bone of the amputated limb. A removable external prosthesis will then be connected to the implant section that protrudes from the soft parts.

The benefits of using an osseointegrated prosthesis are the improved sensory feedback (osseoperception) and absence of the socket. This leads to better anchoring of the prosthesis to the abutment, greater control of the prosthesis and the absence of heat, pain, and pressure sores.

The osseointegrated prosthesis does not reduce the mobility of the limb and promotes good growth of bone and muscle mass. The aim of this study is to evaluate the stability of the osseointegrated implant in trans-femoral and trans-humeral amputees.

The main outcome: quantitative evaluation (rotations, translation and MTPM) of the stability of the implant bone interface by Roentgen Stereo-photogrammetric Analysis (RSA) and follow-up.

The secondary outcome: evaluation of the quality of life improvement in patients through clinical score and satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* BMI<35 kg/m2
* Problem in using socket

Exclusion Criteria:

* Diabetes;
* Peripheral vascular diseases;
* Psychiatric problems;
* Pregnancy;
* Rheumatoid arthritis;
* Neurovascular diseases;
* Neurological deficits;
* Amputation of the contralateral limb;
* Infections in progress;
* Immunosuppression;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Rotation | 24 months
  Rotations X, Y, Z (in degrees) of the implant with respect to the bone
Translation | 24 months
  Translations X, Y, Z (in mm) of the implant with respect to the bone

SECONDARY OUTCOMES:
Health-related quality of life | 24 months
  36-Item Short Form Survey (SF36 )
Pain evaluation | 24 months
  Visual Analog Scale (VAS)
Lower limb: Autonomy | 24 months
  Barthel Index
lower limb: Mobility | 4 months
  Rivermead Mobility Index
Upper limb: functionality | 24 months
  The Disabilities of the Arm, Shoulder and Hand (DASH)
Upper Limb: Development and evaluation of the activities measure for upper limb amputees | 24 months
  Activities Measure for Upper Limb Amputees (AM-ULA)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided